CLINICAL TRIAL: NCT03211078
Title: The Application of Electro-magnetic Navigation Bronchoscopy (ENB) and Photodynamic Therapy in the Treatment for Early Lung Cancer
Brief Title: ENB and Photodynamic Therapy in the Treatment for Early Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201407063DINB
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Lung Cancer
Keywords: Early lung cancer; Photodynamic therapy; ENB
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- super-D ENB guided-PDT (Experimental): To test the feasibility of super-D ENB guided-PDT to treat small lung cancer which cannot be eradicated through surgical resection.
  Interventions: Procedure: super-D ENB guided-PDT

INTERVENTIONS:
Procedure: super-D ENB guided-PDT — PDT with super-D EBN localization will be given for treating the target lung lesion. Intrvenous photofrin (2mg/kg) will be given 48 hours before intervention. After localization of the tumor by ENB, a 630nm of light will be give for the lesion with the dosage of 2oo J/cm. Intravenous general anesthesia and endobronchial intubation will be performed under the whole procedure.

SUMMARY:
With the increased incidence of lung cancer and prevalence of low dose CT screening, treating of early lung cancer has becoming an important issue in the clinical practice of thoracic oncology. In this clinical study, the investigators will evaluate whether superDimension (superD) ENB (Electromagnetic navigation bronchoscopy) in combination with interstitial photodynamic therapy can provide the chance of tumor eradication.

DETAILED DESCRIPTION:
Lung cancer is the one the major cause of cancer death all over the world especially in Asia. The prevalence of low dose CT screening has made more patients of lung cancer treated in the early stage. The treatment of choice for of early lung cancer is surgical resection. However, several difficulties exist in surgery for treating early lung cancer. eg. Some presenting as multi-focal lesions, which cannot be completely eradicated by surgical resection.

Electromagnetic navigation bronchoscopy (ENB)（superDimension™ Navigation System, super-D ENB) is a novel technique, which uses an image guided localization system to direct steerable bronchoscopic tools to predetermined points within the bronchial tree. This technology allows improved access to peripheral lesions in particular.

Photodynamic therapy (PDT) has been adopted an effective treatment option for the central located lung cancer by using photosensitizer which is focally retained in the tumor leading to tumor-specific abrasion by irradiating with a certain wave-length of light. The most frequently used and commercially available photosensitizer for lung cancer is PDT with Photofrin under 623 nm red light irradiation. For the peripheral lung cancer which cannot be approached by bronchoscopy, interstitial PDT with the aids of CT guided catheter implantation has been adopted. However, there are potential disadvantages of such approach including 1) bleeding or hemothorax during CT-guided catheter implantation; 2) dislodging of the catheter after lung collapse in the procedure; 3) unable to treat other lesion after pneumothorax.

In the current proposal, the investigators use ENB in combination with PDT to handle to test the feasibility of super-D ENB guided-PDT to treat small lung cancer which cannot be eradicated through surgical resection.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple small lung cancer which cannot be completely removed by surgical resection.
2. Patient with small early lung cancer with diameter less than 1 cm and with high surgical risk precluding surgery.
3. Patient with small early lung cancer with diameter less than 1 cm but unwilling to receive surgical intervention.
4. Age above 20 years old and who can do the bronchoscopy test

Exclusion Criteria:

1. Bleeding tendency. 2 .Poor cardiopulmonary function with intolerance to bronchoscopy examination.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-09-15 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5 years
  The time interval between enrollment and the earliest onset of any of the following events,: tumor local recurrence , distant metastasis, and mortality

SECONDARY OUTCOMES:
post-operative complication | 3 month
  defined as any deviation from the normal postoperative course
post-operative pulmonary function | 6, 12, and 24 months
  the pulmonary function at 6, 12, and 24 months post-operation
overall survival | 5 years
  The time interval between enrollment and death

CONTACTS AND LOCATIONS:
Overall Officials: Jang-Ming Lee, MD. PhD., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist., Taiwan